CLINICAL TRIAL: NCT07055347
Title: Feasibility Study of Home Cardiac Rehabilitation Program for Postoperative Children With Congenital Heart Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Wei XIA, PhD, Association Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: LSLL2024-801-2
Record Dates: First submitted 2025-06-21; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Congenital Heart Disease (CHD); Preschool Children; Rehabilitation
Keywords: Congenital Heart Disease; preschool children; Postoperative heart rehabilitation; Home rehabilitation
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Home-based cardiac rehabilitation group (Experimental): Participants in this arm will receive a structured home-based cardiac rehabilitation program designed for preschool children (aged 3-7 years) who have undergone corrective surgery for congenital heart disease. The program includes modules on physical activity, breathing exercises, emotional support, and caregiver education. Caregivers will implement the 12-week intervention at home with support materials and guidance provided by the research team.
  Interventions: Other: Comprehensive Home-based Cardiac Rehabilitation Program for Postoperative Congenital Heart Disease Patients and Their Caregivers

INTERVENTIONS:
Other: Comprehensive Home-based Cardiac Rehabilitation Program for Postoperative Congenital Heart Disease Patients and Their Caregivers — Intervention Description: For children, provide age-appropriate rehab manuals with pictures and texts to encourage participation. Include gentle physical activities, breathing and stretching exercises. For caregivers, offer detailed manuals and checklists. Organize training. Manage drugs with personalized guidance. Provide health education for both via manuals and video consultations. Focus on mental and physical health with support and activities. Regular phone follow-ups ensure nursing continuity. Multidisciplinary team offers professional support through video consultations and referrals.

SUMMARY:
This single-arm feasibility study will pilot a home-based cardiac rehabilitation program for preschool children (aged 3 to 7 years) who have undergone corrective surgery for congenital heart disease. Following the development of the program through expert consensus, this phase will implement the preliminary version of the program in a selected sample of caregiver-child pairs over a 12-week period. The study will assess feasibility by evaluating caregiver adherence to the intervention, acceptability of the program components, and completeness of rehabilitation task records. Descriptive data on safety, participation rate, and delivery logistics will also be collected. Findings will inform refinement of the program prior to future effectiveness testing.

ELIGIBILITY:
Children With Congenital Heart Disease After Surgery

Inclusion Criteria:

* Meet the diagnostic criteria for congenital heart disease
* Aged between 3 and 7 years
* Underwent open-heart congenital heart disease correction surgery at the research institution and achieved correction in a single surgery
* Have been discharged after completing inpatient postoperative rehabilitation
* Able to communicate in Chinese

Exclusion Criteria:

* Postoperative arrhythmia
* Neurological, respiratory, or other comorbid diseases in addition to congenital heart disease and assessed by a physician as unsuitable for exercise
* Cardiac function classified as NYHA Class IV
* Intellectual, language, or motor impairments resulting from perioperative complications or other causes

Caregivers of Children With Congenital Heart Disease After Surgery

Inclusion Criteria:

* The primary caregiver of the child, limited to the child's father or mother
* Among parents, the one who has provided care for the longest duration
* Able to communicate in Chinese

Exclusion Criteria:

* Caregivers of children who voluntarily discontinued treatment before its completion
* Paid or non-parental caregivers
* Individuals with diagnosed cognitive impairment or mental illness
* Inability to communicate effectively through spoken language
* Serious conflict or instability in the caregiver-child relationship
* Inability to independently operate and use smart electronic devices and internet-based tools

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Caregiver Adherence Rate to the Home Rehabilitation Program | Up to 4 weeks post-enrollment (exact duration to be finalized)
  During the pilot implementation phase of the home-based rehabilitation program, caregivers will be asked to assist their children in completing assigned daily tasks (e.g., physical activities, breathing exercises, emotional support). Adherence will be tracked using daily caregiver logs. The outcome will be calculated as the percentage of completed tasks over the total assigned tasks per participant. Summary statistics (mean ± SD) will be reported.

SECONDARY OUTCOMES:
Rehabilitation Program Data | At 7 and 14 days after implementation
  collect rehabilitation indicators from caregivers in the form of photos (resting heart rate, heart rate during exercise, Borg's perceived exertion score before and after exercise, complexion, lip color, child's complaint).
Feedback survey | At 7 and 14 days after implementation
  Collect feedback on the trial of the rehabilitation program from caregivers and some older children via phone or online video conference. Focus on collecting compliance-related indicators (e.g., whether rehabilitation training items are completed on time and as required, whether relevant drugs are taken at the prescribed dose, etc.) and acceptability-related indicators (e.g., acceptance of rehabilitation training intensity, methods, duration, etc.).

IPD SHARING:
Plan to Share IPD: No